CLINICAL TRIAL: NCT01518764
Title: The Effects of Red Wine Polyphenols on Microvascular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Erik Serne, MD phd, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL37147.029.11
Record Dates: First submitted 2012-01-02; First posted 2012-01-26 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Red Wine Polyphenols (Experimental): Red Wine Polyphenols 600mg/day (capsules)
  Interventions: Dietary Supplement: Red Wine Polyphenols 600mg/day
- placebo (Placebo Comparator): placebo (capsules)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Red Wine Polyphenols 600mg/day
  Other Names: Provinols™
  Arms: Red Wine Polyphenols
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
Rationale:

Epidemiological studies have shown that consumption of alcoholic beverages, red wine in particular, is associated with less cardiovascular mortality. In addition, there are reported beneficial effects of red wine on components of the metabolic syndrome, arguably the most menacing cardiometabolic condition facing us due to the unfolding obesity epidemic. Beneficial effects have also been reported with other polyphenol-rich food stuff, such as cocoa and green tea and points to a beneficial effect which does not seem to be dependent on the alcohol content of red wine. Experimental studies with mixed or separate Red Wine Polyphenols (RWPs) (i.e. without alcohol) have shown beneficial effects on cardiometabolic parameters associated with obesity. Most research has focused on resveratrol, a specific polyphenol components which is quite specific to red wine and has, at least in animal studies, beneficial effects on insulin sensitivity, insulin secretion, and endothelial function. Moreover, RWPs have shown to improve endothelial NO-mediated relaxation using the same PI3-kinase/Akt pathway as does insulin. However, data in humans are remarkably scarce

Objective:

To study effects of RWPs on insulin sensitivity, beta-cell function, microvascular function (skin, muscle and cardiac), blood pressure, insulin-mediated microvascular responsiveness.

Study design:

Randomized controlled trial (double blind).

Study population:

Obese (BMI >30); n=30, men or women, aged 18-60 years.

Intervention:

Mixed RWP 600mg/day or matching placebo for a total duration of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* age 18-60 years
* obese (BMI >30)

Exclusion Criteria:

* cardiovascular disease
* smoking
* diabetes mellitus
* recent history (<12 months) of high alcohol use > 4 U/day
* use of medication potentially affection insulin sensitivity or microvascular function
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2012-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity as determined by euglycemic clamp tests | 8 weeks

SECONDARY OUTCOMES:
Molecular mechanisms in muscle tissue | 8 weeks
Glucose tolerance as assessed by the area under the curve for glucose (AUCgluc) during a standardized meal test | 8 weeks
microvascular function (baseline and during hyperglycemia) | 8 weeks
Blood pressure 24 hr measurement | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erik Serne, MD PhD, Principal Investigator — VUmc, internal medicine
Locations (1):
- VUMedicalCenter, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Woerdeman J, Del Rio D, Calani L, Eringa EC, Smulders YM, Serne EH. Red wine polyphenols do not improve obesity-associated insulin resistance: A randomized controlled trial. Diabetes Obes Metab. 2018 Jan;20(1):206-210. doi: 10.1111/dom.13044. Epub 2017 Aug 14. PMID 28643477